CLINICAL TRIAL: NCT04171323
Title: ACTIVE MIND: An Adaptive Clinical Trial of Cognitive Training to Improve Function and Delay Dementia
Brief Title: The Active Mind Trial: An Adaptive Randomized Trial to Improve Function and Delay Dementia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Florida (Other); University of Minnesota (Other); National Institute on Aging (NIA) (NIH); Clemson University (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Jerri Edwards, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: WIRB® Protocol #20192632; R01AG075014 (NIH)
Record Dates: First submitted 2019-11-07; First posted 2019-11-20 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Age-related Cognitive Decline; Mild Cognitive Impairment; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CTa (Experimental): Participants will complete computerized cognitive training. The duration is 60 min/day; the frequency is two to three days/wk, for 16 weeks with the goal of completing 40 sessions.
  Interventions: Behavioral: Cognitive Training
- CTab (Experimental): Participants will complete computerized cognitive training. The duration is 60 min/day; the frequency is two to three days/wk, for 16 weeks with the goal of completing 40 sessions.
  Interventions: Behavioral: Cognitive Training
- CTac (Experimental): Participants will complete computerized cognitive training. The duration is 60 min/day; the frequency is two to three days/wk, for 16 weeks with the goal of completing 40 sessions.
  Interventions: Behavioral: Cognitive Training
- CTabc (Experimental): Participants will complete computerized cognitive training. The duration is 60 min/day; the frequency is two to three days/wk, for 16 weeks with the goal of completing 40 sessions.
  Interventions: Behavioral: Cognitive Training
- Computerized Cognitive Stimulation (Active Comparator): Participants will complete cognitively-stimulating computer activities. The duration is 60 min/day; the frequency is two to three days/wk, for 16 weeks with the goal of completing 40 sessions.
  Interventions: Behavioral: Computerized Cognitive Stimulation

INTERVENTIONS:
Behavioral: Cognitive Training — Participants will be completing a total of 40 computerized sessions.
  Arms: CTa; CTab; CTabc; CTac
Behavioral: Computerized Cognitive Stimulation — Participants will be completing a total of 40 computerized cognitive stimulation sessions.
  Arms: Computerized Cognitive Stimulation

SUMMARY:
Older adults at risk for dementia show a variety of cognitive deficits, which can be ameliorated by different cognitive training (CT) exercises. The best combination of CT exercises is unknown. The aim is to discover the most efficacious combination of CT exercises as compared to cognitive stimulation (which will serve as a stringent, active control) to modify the functional trajectories of older adults' with MCI, who are at high risk for dementia. The primary objective of the U01 phase was to design and pilot-test an adaptive, randomized clinical trial (RCT) of cognitive training (CT) combinations aimed to enhance performance of instrumental activities of daily living (IADL) among persons with mild cognitive impairment (MCI). In the R01 phase, the objective is to identify the best combination of CT exercises to delay dementia onset among persons with MCI. The longitudinal endpoint goal is reducing incident dementia. The primary aim of the study is to determine which CT combination has the best probability to delay dementia by producing the largest IADL improvements. The study further aims to explore neuroimaging and novel blood-based biomarkers.

DETAILED DESCRIPTION:
An Adaptive Clinical Trial of Cognitive Training to Improve Function and Delay Dementia: The ACTIVE MIND Trial.

In the U01 phase, the primary objective was to design and pilot-test an adaptive, randomized clinical trial (RCT) of cognitive training (CT) combinations aimed to enhance performance of instrumental activities of daily living (IADL) among persons with mild cognitive impairment (MCI). The longitudinal endpoint goal is delaying dementia onset.

The secondary objectives of the U01 phase were:

- To pilot test a plan to recruit and enroll under-represented minorities with the goal of obtaining a sample representative of the USF population in race and ethnicity.

In the current R01 phase:

The primary objective is to conduct an adaptive, randomized clinical trial (RCT) of cognitive training (CT) combinations aimed to enhance performance of instrumental activities of daily living (IADL) among persons with mild cognitive impairment (MCI). The longitudinal endpoint goal is reducing dementia incidence.

Design: The design is an adaptive randomized trial to identify the best combination of CT exercises to improve IADL function and thereby delay dementia onset among persons with MCI. Four arms of CT will be compared to an active control condition.

Outcomes: incident dementia is the primary outcome. Secondary outcome is Everyday Function: measures include Timed Instrumental Activities of Daily Living and iFunction. A composite of performance (measured by time and accuracy) will be derived.

Interventions and Duration: Four combinations of computerized cognitive training and an active control computerized stimulation will be investigated. The five arms will be equivalent in terms of frequency and duration of each session (60 min/day, two-three days/wk, 16 weeks).

Sample size: The study team plans to enroll up to 1305 participants. Individuals with a clinical diagnosis of MCI will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* 55 to 89 years of age
* Montreal Cognitive Assessment Score of 18-27 inclusive
* History of some change in cognitive function relative to established baseline and either 1) a CDR of 0.5; or 2) CDR of 0 and a clinical diagnosis of mild cognitive impairment (MCI) based on a multidisciplinary evaluation that included standardized neuropsychological testing
* If reports use of medications typically prescribed for dementia such as Namenda, Memantine, Namzaric, Donepezil, Aricept, Rivastigmine, Exelon, Razadyne, Galantamine, or Reminyl, dose has been stable for at least 30 days
* Adequate auditory capacity to understand normal speech. No greater than moderate hearing loss evident by thresholds less than or equal to 50 dB at 1000 and 2000 Hz in at least one ear determined by an audioscope.
* Adequate visual capacity to read from a computer screen at a normal viewing distance as measured by binocular visual acuity of 20/50 or better tested with a standard near visual acuity chart
* Reports and shows adequate motor capacity to touch a computer screen or control a computer mouse.
* Wiling to complete all study activities
* Willing and capable of providing informed consent
* Ability to understand study procedures and comply with them for the length of the study

Exclusion Criteria:

* Currently enrolled in another randomized clinical trial, treatment trial, or another research study that assesses cognition
* Dementia diagnosis
* Clinical Dementia Rating Scale of 1 or greater
* History of large vessel stroke with significant residual motor or cognitive impairment
* History of moderate to severe traumatic brain injury with residual cognitive symptoms
* History of brain tumor
* Undergoing or plans to undergo surgery requiring anesthesia, chemotherapy, or radiation treatment in the six months following screening
* Congestive heart failure diagnosis
* Primary diagnosis of idiopathic Parkinson's disease
* Multiple sclerosis or Amyotrophic lateral sclerosis (ALS) diagnosis
* Evidence of a non-neurodegenerative neurological disorder that would interfere with the ability to carry out study activities.
* Evidence of any other unstable medical conditions that would interfere with the ability to carry out study activities or cause fluctuations in cognition (e.g., unstable diabetes, chronic obstructive pulmonary disorder dependent on oxygen)
* Geriatric Depression short scale score >5/15. Participants with mood disorders that are treated and stable and have a GDS score < 6/15 are not excluded.
* Any other clinically significant or unstable medical condition (e.g., ongoing alcohol dependency or drug abuse, schizophrenia, psychosis) that in the assessor's opinion would interfere with the ability to carry out study activities.
* Previous participation in 10 or more hours of a computerized cognitive intervention program in the past two years
* Previous participation in cognitive intervention research at the study site in the past 2 years
* Planning on going away or being otherwise unavailable for a period of more than three weeks in the six months following screening
* Contraindications to MRI such as pacemaker, metal implants in body, or claustrophobia

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1305 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Dementia incidence | At follow-up visit between 6 months to 2 years
  Clinical diagnosis of dementia

SECONDARY OUTCOMES:
Useful Field of View Test performance overall score | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  Useful Field of View test (UFOV) score across three subtests measured in milliseconds (ms). Lower scores are better.
Graduated continuous performance test score | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  The metrics of performance are target accuracy (in percent correct) and the variability of responses (standard deviation of response times to target images). Higher scores are better.
Examiner Executive Function Set shifting, Anti-Saccades, and Flanker performance composite score | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  The proprietary software calculates an overall executive function composite score using item response theory. Higher scores are better
Timed IADL performance score | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  A composite z score is calculated that reflects the overall time and accuracy of performance on the Timed IADL subtests per standard, published procedures (SPSS syntax of scoring method can be provided). Lower scores are better.
ifunction performance efficiency index | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  An overall score reflecting time and accuracy (i.e., efficiency index) is calculated to reflect performance across the ifunction subtests the proprietary software determines the score. Higher scores are better for efficiency index

OTHER OUTCOMES:
blood based biomarker Neurofilament light (Nfl) | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  Effect sizes of between group differences will be calculated using linear contrasts.
blood based biomarker Total tau | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  Effect sizes of between group differences will be calculated using linear contrast
blood based biomarker hydroxsphingomyelins SM (OH) C22:1, SM (OH) C22:2, SM (OH) C24:1 | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  Effect sizes of between group differences will be calculated using linear contrasts.
blood based biomarker brain derived neurotropic factor (BDNF) | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  Effect sizes of between group differences will be calculated using linear contrasts.
blood based biomarker insulin growth factor-1 (IGF-1), IGF binding protein-1 (IGFBP1) and IGFBP-2 | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  Effect sizes of between group differences will be calculated using linear contrasts.
blood based vascular biomarkers of asymmetric dimethylarginine [ADMA]; aspartic avid; acetyl-L-cartinine [C2]; butenyl-L-cartinine [C4:1] | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  Effect sizes of between group differences will be calculated using linear contrasts.
Neuroimaging MRI whole brain and regional volume | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  Effect sizes of between group differences will be calculated using linear contrasts.
Neuroimaging MRI surface area cortical thickness metrics from T1 weighted images | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  Effect sizes of between group differences will be calculated using linear contrasts.
Neuroimaging MRI whole brain and regional white matter hyper-intensity volume from FLAIR | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  Effect sizes of between group differences will be calculated using linear contrasts.
Neuroimaging MRI hippocampal subfield volume from high resolution hippocampal images | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  Effect sizes of between group differences will be calculated using linear contrasts.
Neuroimaging MRI regional and white matter metrics of fractional anisotropy from diffusion weighted imaging | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  Effect sizes of between group differences will be calculated using linear contrasts.
Neuroimaging MRI regional and white matter metrics of median diffusivity from diffusion weighted imaging | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  Effect sizes of between group differences will be calculated using linear contrasts.
Neuroimaging MRI regional and white matter metrics of radial diffusivity from diffusion weighted imaging | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  Effect sizes of between group differences will be calculated using linear contrasts.
Neuroimaging MRI regional and whole brain measures of cerebral perfusion from arterial spin labeling | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  Effect sizes of between group differences will be calculated using linear contrasts.
Neuroimaging MRI regional and whole brain cerebral microbleed volume from T2*GRE images | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  Effect sizes of between group differences will be calculated using linear contrasts.
Neuroimaging regional and network measures of functional connectivity for resting state fMRI | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  Effect sizes of between group differences will be calculated using linear contrasts.
Virtual Reality Functional Assessment Tool performance | change from baseline to immediate post intervention at the end of study completion which is a period of about 6 months
  Measures may include Virtual Reality Functional Assessment Tool (VRFCAT) Effect sizes of between group differences will be calculated using linear contrasts.

CONTACTS AND LOCATIONS:
Overall Officials: Jerri Edwards, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (6):
- United States (6):
  - University of California San Francisco, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Active Mind Study, Tampa, Florida
  - University of Minnesota, Minneapolis, Minnesota
  - Clemson University, Greenville, South Carolina
  - Clemson University, Seneca, South Carolina